CLINICAL TRIAL: NCT03390244
Title: Foldable Capsular Vitreous Body Implantation Study
Acronym: FCVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Stalmans, Head of Clinic, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S59809
Record Dates: First submitted 2016-12-08; First posted 2018-01-04 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Vitreoretinal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCVB Implant (Experimental): All subjects in this study are in the experimental treatment arm and will receive the FCVB implant
  Interventions: Device: Foldable Capsular Vitreous Body Implant

INTERVENTIONS:
Device: Foldable Capsular Vitreous Body Implant — Vitrectomy augmented with the implantation of the FCVB implant

SUMMARY:
This study is intended to evaluate the clinical usefulness of the FCVB in its on-label use, but in a different racial type than studies till now (Asians only). The device will be inserted in Caucasian patients with permanent loss of functional vision (visual acuity hand movements or less), where a permanent use of repeat silicone oil is required to maintain the eye pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* Axial length between 16 and 28 mm (according the guidelines from the manufacturer)
* Loss of functional vision in study eye
* Visual acuity of 0.4 or better in fellow eye
* Requirement of (repeated) long-term silicone oil tamponade to maintain eye pressure and keep the retina attached

Exclusion Criteria:

* Visual acuity beyond 0.4 in non-study eye
* Severe general disease that is evaluated to impact live expectancy beyond the duration of the study follow-up (3 years)
* Retinal detachment under silicone oil fill
* Patients with a silica gel allergy or scar diathesis
* Patients with serious heart, lung, liver, or kidney dysfunction
* Patients with proliferative diabetic retinopathy, endophthalmia, uveitis and other uncontrollable eye diseases, or a contralateral eye that had intraocular retinal surgery
* Patients with history of drug abuse or alcoholism
* Patients are had participating in other drug or medical device clinical trials before screening for this trial
* Pregnancy, preparation for pregnancy during clinical trial, or breast-feeding
* Belief by any of the research doctors that a patient's condition would hinder the clinical trial, such as a patient prone to mental stress, loss of control of mood, or depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Intra-ocular pressure | 3 years
  Evaluation of the device as long-term solution for maintenance the intra-ocular pressure, potentially reducing the number of surgeries (silicone oil exchanges) for the patient

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, MD Phd, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven (UZLeuven), Leuven, Vl-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No